CLINICAL TRIAL: NCT05234554
Title: The INVIGORATE 2 Trial: A Single-center, Randomized, Double-masked, Crossover Design, Vehicle-controlled, Phase 3 Clinical Trial to Assess the Efficacy and Safety of Reproxalap Ophthalmic Solution (0.25%) Compared to Vehicle in Subjects With Seasonal Allergic Conjunctivitis Using the Environmental Exposure Chamber (EEC)
Brief Title: The INVIGORATE 2 Trial: A Clinical Trial to Assess the Efficacy and Safety of Subjects With Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADX-102-AC-026
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) dosed twice.
  Arms: Reproxalap Ophthalmic Solution (0.25%)
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution dosed twice.
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
The INVIGORATE 2 Trial: A single-center, randomized, double-masked, crossover design, vehicle-controlled, Phase 3 clinical trial to assess the efficacy and safety of reproxalap ophthalmic solution (0.25%) compared to vehicle in subjects with seasonal allergic conjunctivitis using the environmental exposure chamber (EEC).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at the time of screening of either sex or any race;
* Provide written informed consent;
* Be willing and able to follow instructions, and can attend all required clinical trial visits.
* Have at least a two-year history of moderate-to-severe ragweed-induced allergic conjunctivitis based on investigator's judgement;
* Have a positive skin prick test to ragweed pollen within the past year of the Medical Screening Visit (Visit 1).

Exclusion Criteria:

* Have a history of blepharitis, dry eye syndrome, herpes simplex keratitis, or herpes zoster keratitis;
* Have systemic signs of infection (e.g., fever, current treatment with antibiotics).
* Have a systemic disease or uncontrolled medical condition, which, in the opinion of the investigator, could interfere with clinical trial measurements or subject compliance. Such diseases or conditions would include, but are not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease;
* Be a WOCBP who is pregnant, nursing, or not using an effective means of contraception;
* Have any known contraindication or hypersensitivities to any components of the Investigational Product (IP) drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Ocular itching evaluated by the Subject. | During EEC allergen exposure.
  The method of assessment for the primary outcome is a 9-point ocular itch scale (0 none - 4 severe).

SECONDARY OUTCOMES:
Conjunctival redness evaluated by the Subject. | During EEC allergen exposure.
  The method of assessment for the key secondary outcome is a 9-point ocular redness scale (0 none - 4 extremely severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No